CLINICAL TRIAL: NCT00765999
Title: An Open-Label, Long-Term Safety Study of Oral Linaclotide Administered to Patients With Chronic Constipation or Irritable Bowel Syndrome With Constipation
Brief Title: An Open-Label, Long-Term Safety Study of Linaclotide in Patients With Chronic Constipation or Irritable Bowel Syndrome With Constipation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Ironwood Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LIN-MD-02
Record Dates: First submitted 2008-10-01; First posted 2008-10-03 (Estimated); Results first posted 2019-02-15 (Actual); Last update posted 2019-02-15 (Actual); Status verified 2019-01

CONDITIONS: Chronic Constipation; Irritable Bowel Syndrome With Constipation
Keywords: Constipation; Chronic Constipation; Irritable Bowel Syndrome With Constipation; Linaclotide
MeSH Terms: conditions — Constipation | interventions — linaclotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Linaclotide (Experimental): Linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks in participants with either CC or IBS-C. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced AEs intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, participants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
  Interventions: Drug: Linaclotide

INTERVENTIONS:
Drug: Linaclotide — Linaclotide capsules, oral, once daily each morning at least 30 minutes before breakfast for the duration of the study.
  Other Names: Linzess

SUMMARY:
The objective of this study is to assess the long-term safety of linaclotide administered to patients with chronic constipation (CC) or irritable bowel syndrome with constipation (IBS-C).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have

  * entered study LIN-MD 01[NCT00765882] or LIN-MD-31 [NCT00948818] and at minimum completed the pre-treatment period or
  * completed one of the following studies: MCP-103-004 [NCT00306748], MCP-103-005 [NCT00258193], MCP-103-201 [NCT00402337], MCP-103-202 [NCT00460811]
* Sexually active patients of childbearing potential agree to use birth control
* Females of childbearing potential must have a negative urine pregnancy test prior to dosing
* Lactating females must agree not to breastfeed
* Patient must meet protocol criteria for CC or IBS-C

Exclusion Criteria:

* Patient must not use protocol-defined prohibited medicine
* Patient is planning to receive an investigational drug at any time during the study
* Patient has an unresolved AE or a clinically significant finding on a physical examination, 12-lead ECG, or clinical laboratory test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1559 (Actual)
Dates: Start 2008-10-31 (Actual); Primary Completion 2012-01-31 (Actual); Study Completion 2012-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Eng, PhD, Study Director — Forest Laboratories
Locations (117):
- United States (109):
  - Innovative Clinical Trials, Birmingham, Alabama
  - Parkway Medical Center, Birmingham, Alabama
  - Medical Affiliated Research Center, Inc., Huntsville, Alabama
  - Radiant Research, Inc., Chandler, Arizona
  - Pivotal Research Centers, Peoria, Arizona
  - Pivotal Research Center, Peoria, Arizona
  - Carl T Hayden VA Medical Center GI Section-CS-111G, Phoenix, Arizona
  - Elite Clinical Studies, LLC, Phoenix, Arizona
  - Radiant Research, Inc., Scottsdale, Arizona
  - Genova Clinical Research, Inc., Tucson, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Providence Clinical Research, Burbank, California
  - Encompass Clinical Research North Coast, Encinitas, California
  - Family Medical Center, Foothill Ranch, California
  - Axis Clinical Trials, Los Angeles, California
  - Facey Medical Foundation, Mission Hills, California
  - Advanced Clinical Research Institute, Orange, California
  - Westlake Medical Research, Westlake Village, California
  - Boulder Medical Center, P.C., Boulder, Colorado
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Colorado Gastroenterology, Prof LLC, Denver, Colorado
  - Longmont Medical Research Network, Longmont, Colorado
  - Western States Clinical Research, Wheat Ridge, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Clinical Trials Management of Boca Raton, Inc., Boca Raton, Florida
  - Meridien Research, Bradenton, Florida
  - PAB Clinical Research, Brandon, Florida
  - Meridien Research, Brooksville, Florida
  - Clinical Physiology Associates Clinical Study Center, Fort Myers, Florida
  - Jupiter Research, Inc., Jupiter, Florida
  - FPA Clinical Research, Kissimmee, Florida
  - Pharmax Research Clinic, Miami, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - RenStar Medical Research, Ocala, Florida
  - Compass Research, Orlando, Florida
  - Emerald Coast Research Associates, Panama City, Florida
  - University Clinical Research, Inc., Pembroke Pines, Florida
  - Miami Research Associates, South Miami, Florida
  - Meridien Research, St. Petersburg, Florida
  - Meridien Research, Tampa, Florida
  - Advanced Research Institute, Trinity, Florida
  - Florida Medical Clinic, P.A. Clinical Research Division, Zephyrhills, Florida
  - Radiant Research, Inc., Atlanta, Georgia
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Atlanta Gastroenterology Associates, LLC, Marietta, Georgia
  - Clinical Research Atlanta, Stockbridge, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - Rosemark WomenCare Specialist, Idaho Falls, Idaho
  - Rockford Gastroenterology Associates, Ltd., Rockford, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Heartland Research Associates, LLC, Arkansas City, Kansas
  - Heartland Research Associates, LLC, Newton, Kansas
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Central Kentucky Research Associates, Lexington, Kentucky
  - Trover Health System, Madisonville, Kentucky
  - Medical Development Centers, LLC, Baton Rouge, Louisiana
  - Clinical Trials of America, Inc., Shreveport, Louisiana
  - Metropolitan Gastroenterology Group PC, Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Meritus Center for Clinical Research, Hagerstown, Maryland
  - Charm City Research, Towson, Maryland
  - Boston Clinical Trials, Boston, Massachusetts
  - Kalamazoo Gastroenterology Hepatology, Kalamazoo, Michigan
  - Ridgeview Research Two Twelve Medical Center, Chaska, Minnesota
  - St. Louis Center for Clinical Research, St Louis, Missouri
  - The Gastroenterology Group of S.J., Vineland, New Jersey
  - New Mexico Clinical Research and Osteoporosis Center, Albuquerque, New Mexico
  - Lifeline Research Institute, Brooklyn, New York
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Long Island Gastrointestinal Research Group, Great Neck, New York
  - Gastrointestinal Research Associates, LLC, Setauket, New York
  - MediSpect, LLC, Boone, North Carolina
  - Cumberland Research Associates, LLC, Fayetteville, North Carolina
  - LeBauer Research Associates, P.A., Greensboro, North Carolina
  - Clinical Trials of America, INC, Hickory, North Carolina
  - Wake Research Associates, LLC, Raleigh, North Carolina
  - Hanover Medical Specialists, PA, Wilmington, North Carolina
  - Digestive Health Specialists, PA, Winston-Salem, North Carolina
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Remington Davis, Columbus, Ohio
  - Hometown Urgent Care and Research, Dayton, Ohio
  - Oklahoma Foundation for Digestive Research, Oklahoma City, Oklahoma
  - Gastroenterology United of Tulsa, Tulsa, Oklahoma
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - Mountain View Clinical Research, Greer, South Carolina
  - Radiant Research, Greer, South Carolina
  - Nashville Medical Research Institute, Nashville, Tennessee
  - Professional Quality Research, Inc., Austin, Texas
  - Research Across America RHD Professional Plaza IV, Dallas, Texas
  - Houston Digestive Diseases Clinic, Houston, Texas
  - Houston Medical Research Associates, Houston, Texas
  - R/D Clinical Research, Inc., Lake Jackson, Texas
  - Quality Research Inc., San Antonio, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Fatigue Consultation Clinic, Salt Lake City, Utah
  - Department of Gastroenterology University of Utah Hospital, Salt Lake City, Utah
  - Department of Veterans Affairs Research Department, Salt Lake City, Utah
  - Charlottesville Medical Research, Charlottesville, Virginia
  - New River Valley Research Institute, Christiansburg, Virginia
  - Health Research of Hampton Roads, Newport News, Virginia
  - National Clinical Research - Norfolk, Inc., Norfolk, Virginia
  - Clinical Research Associates of Tidewater, Norfolk, Virginia
  - National Clinical Research-Richmond, Inc., Richmond, Virginia
  - Northwest Gastroenterology Associates, Bellevue, Washington
  - Radiant Research, Inc., Lakewood, Washington
  - Wenatchee Valley Medical Center Clinical Research Dept., Wenatchee, Washington
  - Aurora Advanced Healthcare, Inc. Clinical Research Center, Milwaukee, Wisconsin
- Canada (8):
  - GI Research Institute, Vancouver, British Columbia
  - Medicor Research, Inc., Greater Sudbury, Ontario
  - St. Joseph Healthcare, Hamilton, Ontario
  - MedPhase Canada, Newmarket, Ontario
  - Meadowlands Family Health Center, Ottawa, Ontario
  - London Road Diagnostic Clinic and Medical Center, Sarnia, Ontario
  - PrimeHealth Clinical Research, Toronto, Ontario
  - Toronto Digestive Disease Associates, Inc., Vaughan, Ontario

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1559 enrolled participants, all but 5 also received study drug, leading to an overall safety population of 1554 participants.
Groups:
- Linaclotide: Linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks in participants with either CC or IBS-C. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced adverse events (AEs) intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, participants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
Period: Overall Study
Arm/Group | Linaclotide
Started | 1554
Completed | 770
Not Completed | 784
Not completed — Adverse Event | 203
Not completed — Insufficient Therapeutic Response | 100
Not completed — Protocol Violation | 95
Not completed — Consent Withdrawn | 202
Not completed — Lost to Follow-up | 131
Not completed — Study Terminated by Sponsor | 2
Not completed — Other Miscellaneous Reasons | 51

BASELINE CHARACTERISTICS:
Population: Of the 1559 enrolled participants, all but 5 also received study drug, leading to an overall safety population of 1554 participants.
Arm/Group | Linaclotide
Number analyzed (Participants) | 1554
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.0 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1414
  Male | 140
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 1197
  African American | 312
  Other | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic | 192
  Non-Hispanic | 1362
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 76.02 (17.85)
Height [Mean (Standard Deviation); unit: centimeters (cm)] | 164.59 (8.05)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 28.03 (6.14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Treatment-Emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant administered study drug. An AE could, therefore, be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of the study drug, whether or not related to the medicinal product. An AE that occurred during the treatment period was defined as a TEAE if the AE was either not present at, or before, the day of the first dose of open-label study medication in this study or was present at, or before, the day of the first dose of open-label study medication in this study and increased in severity during the treatment period. AEs included abnormal clinically significant findings for clinical laboratory tests, physical examination findings, vital sign measurements and electrocardiograms (ECGs).
Time Frame: Up to 78 weeks for AEs; within 30 days of last dose of study drug (up to 82 weeks) for serious AEs.
Population: The analysis population consisted of participants in the Enrolled Population who received at least 1 dose of the open-label investigational product. It was identified that 1 participant enrolled twice in the study under 2 ID numbers; this participant is included in both the IBS-C and CC Safety Populations, leading to an analyzed population of 1555.
Measure: Count of Participants; unit: Participants
Groups:
- Linaclotide (CC): Linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks in participants with CC. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced AEs intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, paticipants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
- Linaclotide (IBS-C): Linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks in participants with IBS-C. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced AEs intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, participants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
Arm/Group | Linaclotide (CC) | Linaclotide (IBS-C)
Number analyzed (Participants) | 523 | 1032
Participants | 399 | 748

ADVERSE EVENTS:
Time Frame: Up to 78 weeks for AEs; within 30 days of last dose of study drug (up to 82 weeks) for serious AEs.
Description: The safety population consisted of all participants in the Enrolled Population who received at least 1 dose of the open-label investigational product. It was identified that 1 participant enrolled twice in the study under 2 ID numbers; this participant is included in both the IBS-C and CC Safety Populations, leading to an analyzed population of 1555.
Groups:
- Linaclotide (CC): Linaclotide 290 μg/day capsules, administered orally once daily for up to 78 weeks in participants with CC. Dose reduction to 145 μg/day was permitted at the discretion of the Investigator if a participant experienced AEs intolerable enough to prompt consideration of study withdrawal. After a temporary suspension of dosing, participants may have received either 145 μg/day or 290 μg/day of linaclotide, at the discretion of the Investigator. Subsequent dose adjustments (increases or decreases between 290 μg/day and 145 μg/day) were permitted also at the Investigator's discretion.
Arm/Group | Linaclotide (CC) | Linaclotide (IBS-C)
Serious Adverse Events (participants affected / at risk) | 31/523 | 57/1032
Other Adverse Events (participants affected / at risk) | 267/523 | 510/1032
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Linaclotide (CC) (N=523) | Linaclotide (IBS-C) (N=1032)
Cholelithiasis (Hepatobiliary disorders) | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Bladder prolapse (Renal and urinary disorders) | 2 | 0
Cholecystitis (Hepatobiliary disorders) | 2 | 2
Goitre (Endocrine disorders) | 2 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Syncope (Nervous system disorders) | 2 | 2
Uterine prolapse (Reproductive system and breast disorders) | 2 | 0
Abdominal abscess (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Adenomyosis (Reproductive system and breast disorders) | 1 | 1
Angina pectoris (Cardiac disorders) | 1 | 3
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1
Bunion (Surgical and medical procedures) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypertension (Vascular disorders) | 1 | 1
Non-cardiac chest pain (General disorders) | 1 | 4
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 2
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Post procedural infection (Infections and infestations) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Scoliosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spigelian hernia (Gastrointestinal disorders) | 1 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Suicide attempt (Psychiatric disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transient ischaemic attack (Vascular disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Urinary retention postoperative (Injury, poisoning and procedural complications) | 0 | 1
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 | 1
Ventricular tachycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vestibular neuronitis (Infections and infestations) | 0 | 1
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Injury (Injury, poisoning and procedural complications) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Menorrhagia (Reproductive system and breast disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1
Pelvic adhesions (Reproductive system and breast disorders) | 0 | 1
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Stress urinary incontinence (Renal and urinary disorders) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cystocele (Reproductive system and breast disorders) | 0 | 2
Ileus (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Adhesion (General disorders) | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Linaclotide (CC) (N=523) | Linaclotide (IBS-C) (N=1032)
Diarrhoea (Gastrointestinal disorders) | 179 | 345
Abdominal pain (Gastrointestinal disorders) | 34 | 69
Nausea (Gastrointestinal disorders) | 29 | 51
Abdominal distension (Gastrointestinal disorders) | 28 | 35
Upper respiratory tract infection (Infections and infestations) | 31 | 65
Sinusitis (Infections and infestations) | 32 | 61
Urinary tract infection (Infections and infestations) | 30 | 58
Headache (Nervous system disorders) | 34 | 42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor may request the PI delay submission for any publication while the sponsor files applications for patents or other registrations of intellectual property rights.